CLINICAL TRIAL: NCT07121309
Title: Establishment of a Postoperative Delirium Risk Prediction Model for Elderly Hip Fracture Patients Based on Machine Learning Algorithms
Brief Title: With the Development of Research, New Algorithms and Technologies Have Emerged, One of Which is Machine Learning. Machine Learning Can Extract Key Factors From Vast Amounts of Data, Identify Underlying Patterns, and Predict Future Trends. In Recent Years, Machine Learning Has Been Widely Used in
Acronym: POD
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Other Study IDs: JD-HG-2025-022; JD-HG-2025-022 (Other: SecondSoochowU)
Record Dates: First submitted 2025-08-06; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Delirium
Keywords: Hip fracture; Prediction model
MeSH Terms: conditions — Delirium; Hip Fractures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to construct a predictive model for postoperative delirium in elderly patients with hip fractures. The main question it answers is to construct a risk prediction model for hip fractures in the elderly through six machine learning methods, compare which method's model is better, and conduct external validation of the model's stability to provide a reference for the early clinical detection of postoperative delirium in elderly hip fracture patients.

The clinical data of elderly patients with hip fractures have been collected in clinical practice and the model has been constructed.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 60 years; diagnosed with hip fracture by X-ray; patients who underwent surgical treatment.

Exclusion Criteria:

* Patients with other severe diseases (Patients who reach grade IV or higher according to the American Society of Anesthesiologists (ASA) health status classification;Suffer from end-stage diseases;there is multiple organ dysfunction syndrome (MODS) or single organ failure); patients with mental disorders; patients participating in other studies.

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients over 60 years old who undergo surgical treatment for hip fractures
Sampling Method: Probability Sample
Enrollment: 901 (Actual)
Dates: Start 2024-10-17 (Actual); Primary Completion 2025-03-03 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
Postoperative delirium | The day after the operation
  The Memory and Delirium Assessment Scale (MDAS) was used for delirium risk screening and assessment, including consciousness, attention, speech, behavior, and sleep aspects.

CONTACTS AND LOCATIONS:
Locations (1):
- SecondSoochowU, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No